CLINICAL TRIAL: NCT05175001
Title: Efficacy of Compound Betamethasone Injection Combined With Ropivacaine in Ultrasound-guided Thoracic Paravertebral Nerve Block for Chronic Post-thoracotomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Yibin Qin, Associate chief physician, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AHNantongUniversity
Record Dates: First submitted 2021-12-07; First posted 2022-01-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Chronic Pain
Keywords: chronic pain; nerve block
MeSH Terms: conditions — Chronic Pain | interventions — betamethasone dipropionate, betamethasone sodium phosphate drug combination; Ropivacaine

STUDY DESIGN:
Intervention Model Description: The patient is placed in lateral decubitus position with the operative side facing up, and the thoracic paravertebral nerve block will be performed under ultrasound. We select T4-5,T6-7and T8-9 intervertebral spaces for puncture.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: None of the participants know which group they were in,neither of the investigators and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R (Placebo Comparator): The patient is placed in lateral decubitus position with the operative side facing up, and the thoracic paravertebral nerve block will be performed under ultrasound. We select T4-5,T6-7and T8-9 intervertebral spaces for puncture.A 30-mL bolus of a solution of 0.33% ropivacaine in saline was administered under real-time ultrasound monitoring
  Interventions: Drug: Ropivacaine
- Group RD (Experimental): The patient is placed in lateral decubitus position with the operative side facing up, and the thoracic paravertebral nerve block will be performed under ultrasound. We select T4-5,T6-7and T8-9 intervertebral spaces for puncture.A 30-mL bolus of a solution of 0.33% ropivacaine plus 4.67mg Diprospan in saline was administered under real-time ultrasound monitoring
  Interventions: Drug: Diprospan

INTERVENTIONS:
Drug: Diprospan — Diprospan combined with ropivacaine in ultrasound-guided thoracic paravertebral nerve block
  Other Names: Compound Betamethasone Injection
  Arms: Group RD
Drug: Ropivacaine — Only ropivacaine in ultrasound-guided thoracic paravertebral nerve block
  Arms: Group R

SUMMARY:
Chronic post-thoracotomy pain（CPTP）will not only have a negative impact on patients' physiology and psychology, but also affect postoperative recovery.A number of researches have demonstrated that Injury to the intercostal nerve during surgery predominantly accounts for the onset of CPTP.It is closely related to postoperative local acute inflammation and neuroinflammation. Thoracic paravertebral block (TPVB)has become a new trend for post-thoracotomy pain management.Glucocorticoids,as a adjuvant, are reported to prolong the effects of local anesthetic for peripheral nerve blocks.Diprospan is a long-acting glucocorticoid. It has been widely used in clinical treatment of various pain syndromes for powerful analgesic and anti-inflammatory effects. At present, most clinical reports are limited to the acute postoperative period, and there are few studies focusing on the long-term postoperative analgesic effect of diprospan.Therefore, it is reasonable for us to hypothesise diprospan, as a longer-acting glucocorticoid, can provide more lasting analgesic effects,or even reduce the incidence of CPTP

DETAILED DESCRIPTION:
PARAVERTEBRAL BLOCK (PVB) involves the injection of local anesthetic (LA) into a wedge-shaped space lateral to the spinal nerves as they emerge from the intervertebral foramina, producing ipsilateral somatosensory and sympathetic nerve blockade.Since its initial application in abdominal surgery, the technique has been adapted for rib fracture, flflail chest, open cholecystectomy, hepatic-biliary surgery, outpatient inguinal hernia repair, major breast cancer surgery, and open thoracotomy patient populations.Based on several recent systematic reviews and metaanalyses,TPVB and TEA are equal in analgesic effect after thoracic surgery. Moreover, TPVB is associated with fewer side effects,such as urinary retention,nausea/vomiting,pruritus and hypotension. It can also be used for patients with coagulation disorders. Kang et al. argued that TPVB can significantly improve postoperative rehabilitation in patients undergoing thoracoscopic radical lung cancer surgery .

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years
2. American Society of Anesthesiologists(ASA) physical status of I-III
3. BMI: 18.5-28 kg/m2
4. Type of operation: elective thoracoscopic lobectomy
5. The patient and/or family members have signed the informed consent -

Exclusion Criteria:

1. Allergic to local anesthetics or glucocorticoids
2. Preoperative use of opioids
3. Severe coagulation dysfunction
4. Severe heart, lung, liver and kidney insufficiency
5. Used to have immunosuppressive therapies such as radiotherapy, chemotherapy and glucocorticoid, or have immune system diseases
6. Peptic ulcer
7. Perform astrointestinal anastomosis recently
8. Used to have a chest surgery
9. Central nervous system disease or peripheral neuropathy
10. Perioperative blood transfusion
11. Others: such as fracture, wound repair, corneal ulcer, adrenal hypercortical disease, diabetes, pregnant women -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Acute and chronic postoperative pain | 24 hours after surgery
  Numeric rating scale(NRS) is used to assess acute postoperative pain
Acute and chronic postoperative pain | 48 hours after surgery
  Numeric rating scale(NRS) is used to assess acute postoperative pain
Acute and chronic postoperative pain | 72 hours after surgery
  Numeric rating scale(NRS) is used to assess acute postoperative pain
Acute and chronic postoperative pain | 1 month after surgery
  Numeric rating scale(NRS) is used to assess chronic postoperative pain
Acute and chronic postoperative pain | 3 months after surgery
  Numeric rating scale(NRS) is used to assess chronic postoperative pain
Acute and chronic postoperative pain | 6 months after surgery
  Numeric rating scale(NRS) is used to assess chronic postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Yibin Qin, Associate chief physician, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang YK, Yang H, Zhang JY, Song LJ, Fan YC. Comparison of intramuscular compound betamethasone and oral diclofenac sodium in the treatment of acute attacks of gout. Int J Clin Pract. 2014 May;68(5):633-8. doi: 10.1111/ijcp.12359. Epub 2014 Jan 29. PMID 24472084
- [Result] Marty P, Bennis M, Legaillard B, Cavaignac E, Ferre F, Lebon J, Brouchet A, Minville V. A New Step Toward Evidence of In Vivo Perineural Dexamethasone Safety: An Animal Study. Reg Anesth Pain Med. 2018 Feb;43(2):180-185. doi: 10.1097/AAP.0000000000000392. PMID 28394848
- [Result] Watanabe K, Tokumine J, Yorozu T, Moriyama K, Sakamoto H, Inoue T. Particulate-steroid betamethasone added to ropivacaine in interscalene brachial plexus block for arthroscopic rotator cuff repair improves postoperative analgesia. BMC Anesthesiol. 2016 Oct 4;16(1):84. doi: 10.1186/s12871-016-0251-9. PMID 27716229
- [Result] Wang QS, Jiang YH, Wang TD, Xiao T, Wang JK. Effects of betamethasone on neuropathic pain in a rat spare nerve injury model. Clin Exp Pharmacol Physiol. 2013 Jan;40(1):22-7. doi: 10.1111/1440-1681.12027. PMID 23121415